CLINICAL TRIAL: NCT00664885
Title: Effectiveness of Cultural Sensitive Collaborative Treatment of Depressed Chinese in Primary Care
Brief Title: Effectiveness of Cultural Sensitive Collaborative Treatment of Depressed Chinese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Shen-Ing,Liu, Department of Psychiatry, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHRI-EX97-9706PI
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Depression
Keywords: non-psychiatric; clinics
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- CSCT (Experimental)
  Interventions: Other: Culturally Sensitive Collaborative Treatment

INTERVENTIONS:
Other: Culturally Sensitive Collaborative Treatment — a collaborative care model, for treating depressed patients in general medical care

SUMMARY:
This study is a randomized controlled trial to test whether Culturally Sensitive Collaborative Treatment (CSCT) would improve the outcome of depressed patients visiting non-psychiatric settings in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who attend non-psychiatric clinics at the above site.
* Patients with Major Depressive Disorder (MDD), defined as a positive screen using the PHQ-9, confirmed with the SCAN interview.
* Men or women aged 18 or older.
* Able to participate in a clinical diagnostic interview in either Mandarin or Fukienese dialects.
* Individuals who are willing to be followed up concerning their depression symptoms.
* Individuals who have completed a written consent form.

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or planning pregnancy within the next year.
* Patients with serious suicidal risk.
* Patients with unstable medical illnesses.
* Clinical or laboratory evidence of hypothyroidism.
* Patients with comorbid severe mental disorders
* Patients with history of treatment by a psychiatrist in the past 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-01; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Depressed patients who receive CSCT have improved treatment outcomes compared to patients who receive usual care. | 2wk,6 wk,10 wk,14 wk,18 wk,22wk,26wk

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan